CLINICAL TRIAL: NCT02440906
Title: Evaluation of the Texas Wellness Incentives and Navigation (WIN) Project
Acronym: WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); RTI International (Other); Econometrica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 168-2012
Record Dates: First submitted 2015-04-22; First posted 2015-05-12 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Chronic Mental Illness; Chronic Physical Illness
Keywords: Asthma; Cerebrovascular Disease; Intracranial Injury; Neoplasms; Heart Failure; HIV/AIDs; Hereditary and Degenerative Diseases of the Central Nervous System; Disorders of the Peripheral Nervous System; Rheumatoid Arthritis and Other Inflammatory Polyarthropathies; History of hepatitis C; Schizophrenia; Episodic Mood Disorders; Delusional Disorders; Other Non-Organic Psychoses; Organic Psychotic Conditions; Neurotic Disorders; Other Non-Psychotic Mental Disorders
MeSH Terms: conditions — Asthma; Cerebrovascular Disorders; Neoplasms; Heart Failure; Acquired Immunodeficiency Syndrome; Neuritis; Arthritis, Rheumatoid; Schizophrenia; Schizophrenia, Paranoid; Neurotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): A person-centered wellness intervention that includes a patient-directed wellness account. Enrollees meet with a patient Navigator to develop a wellness plan. The enrollee can then use the flexible wellness account to make purchases that are consistent with the goals of the wellness plan. Health Navigators have monthly phone contact with enrollees and meet quarterly with them to discuss goals and spending with the express goal of improving self-management, use of preventive services, satisfaction with care, healthcare utilization and expenditures and quality of care.
  Interventions: Behavioral: Patient-Directed Wellness Account; Behavioral: Health Navigator
- Control (No Intervention): Control group participants receive a monthly mailing requesting updated contact information. They can send this card via mail, or by calling the toll free number.
- Comparison (No Intervention): These are STAR+PLUS enrollees who meet the same enrollment criteria as the intervention and control but reside outside of the Harris Service Area. The purpose of the comparison group is to follow them and their outcomes. This group will help us to better compare the outcomes we see with those enrolled in the WIN Project to a comparable group for whom we already house data.

INTERVENTIONS:
Behavioral: Patient-Directed Wellness Account — The intervention group (n=629) continue to receive usual care and receive a financial incentive to use in meeting their health goals.
  Arms: Intervention
Behavioral: Health Navigator — The intervention group (n=629) will work with a health navigator on a monthly basis to develop and refine patient-centered health goals. Motivational interviewing techniques are used to establish the wellness goals.
  Arms: Intervention

SUMMARY:
The Wellness Incentives and Navigation (WIN) project is designed to help improve health self-management and reduce the incidence and consequences of chronic disease among non-elderly adult Medicaid Supplemental Security Income (SSI) beneficiaries. WIN targets SSI beneficiaries with behavioral health (mental health and substance abuse) diagnoses. Research demonstrates that these individuals are more likely to suffer chronic physical co-morbidities, experience debilitating chronic illnesses earlier in life and have elevated healthcare costs.

WIN uses person-centered wellness planning and navigation facilitated by trained, professional health Navigators, dedicated specifically to the WIN project, who use Motivational Interviewing (MI) techniques, and a personal wellness account. Participants with more serious mental illnesses will be offered additional support in the form of Wellness Recovery Action Planning (WRAP) to enable them to take full advantage of person-centered wellness planning.

DETAILED DESCRIPTION:
The Texas based Wellness Incentives and Navigation (WIN) project uses a continuum of evidence-based "whole person" interventions that take into account clinical, environmental, and social risk factors and co-morbidities. Unlike more traditional didactic approaches to health management, WIN addresses individual behavioral, social, and economic barriers to health and wellness, and promotes continued engagement in achieving, internalizing, and maintaining healthy behaviors.

The study is focused on non-dual eligible adult STAR+PLUS (a Texas Medicaid managed care program for people with chronic illnesses) members (ages 21-55) with a behavioral health disorder including serious mental illness (SMI - e.g., schizophrenia, bipolar disorder or major depressive disorder) or other behavioral health conditions (e.g., anxiety disorder or substance abuse). Key features of the program include the use of professional health navigators, working in collaboration with the three STAR+PLUS plans in the Harris Service Area (SA) (United-Evercare, Amerigroup, and Molina), the use of motivational interviewing (MI) techniques to help members develop and meet personal wellness goals, and a flexible wellness account for the participant to use in meeting his/her goals.

ELIGIBILITY:
Inclusion Criteria:

* Be a resident of the Harris service area
* Be a non-dual eligible member of STAR+PLUS;
* Be 21 to 55 years of age; and
* Have an SMI Diagnosis (schizophrenia, bi-polar disorder, major depressive disorder); or
* Other behavioral health diagnoses (e.g., anxiety, depression, substance use disorder) coupled with a chronic health diagnosis (physical health condition).

Exclusion Criteria:

* Intellectual or cognitive diagnoses indicative of severe cognitive impairment. These could include diagnoses such as 290.X (dementia) and 318-319 (moderate to severe mental retardation).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1663 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Self-reported physical health related quality of life (HRQOL) using the Short Form-12 (SF-12) | (Change) baseline, 12 months, 24 months and 36 months
  The SF-12 has been validated across a number of chronic diseases and conditions. The survey consists of 12 questions measuring functional health and well-being. Patients answer questions related to daily functioning, difficulties in physical tasks, and disruptions in life due to mental illness (e.g. depression, anxiety). The overall score can be further classified into two summary scores for physical and mental health.
Self-reported mental health related quality of life (HRQOL) using the Short Form-12 (SF-12) | (Change) baseline, 12 months, 24 months and 36 months
  The SF-12 has been validated across a number of chronic diseases and conditions. The survey consists of 12 questions measuring functional health and well-being. Patients answer questions related to daily functioning, difficulties in physical tasks, and disruptions in life due to mental illness (e.g. depression, anxiety). The overall score can be further classified into two summary scores for physical and mental health.

SECONDARY OUTCOMES:
Change in Total Healthcare expenditures as measured through Medicaid claims data | (Change) baseline, 12 months, 24 months, 36 months, and 1 year after month 36
  We will use Medicaid claims and enrollment expenditure data to examine changes in total medical expenditures between the three groups of participants across baseline, 12 months, 24 months and 36 months.
Changes in Inpatient Hospitalization expenditures as measured through Medicaid claims data | (Change) baseline, 12 months, 24 months, 36 months, and 1 year after month 36
  We will use Medicaid claims and enrollment expenditure data to examine changes in inpatient hospitalization expenditures between the three groups of participants across baseline, 12 months, 24 months and 36 months.
Changes in Outpatient expenditures as measured through Medicaid claims data | (Change) baseline, 12 months, 24 months, 36 months, and 1 year after month 36
  We will use Medicaid claims and enrollment expenditure data to examine changes in outpatient expenditures between the three groups of participants across baseline, 12 months, 24 months and 36 months.
Changes in Emergency Department expenditures as measured through Medicaid claims data | (Change) baseline, 12 months, 24 months, 36 months, and 1 year after month 36
  We will use Medicaid claims and enrollment expenditure data to examine changes in emergency department expenditures between the three groups of participants across baseline, 12 months, 24 months and 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shenkman, Ph.D., Principal Investigator — University of Florida; Kimberly Case, Ph.D., Study Director — University of Florida; Dena Stoner, Study Director — Texas Health and Human Services Commission
Locations (1):
- University of Florida, Institute for Child Health Policy, Gainesville, Florida, United States

REFERENCES:
- [Derived] Shenkman E, Muller K, Vogel B, Nixon SJ, Wagenaar AC, Case K, Guo Y, Wegman M, Aric J, Stoner D. The wellness incentives and navigation project: design and methods. BMC Health Serv Res. 2015 Dec 29;15:579. doi: 10.1186/s12913-015-1245-x. PMID 26714845